CLINICAL TRIAL: NCT01936480
Title: Genetics of QT Response to Moxifloxacin
Acronym: MOXIGEN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christopher Newton-Cheh, MD, Christopher Newton-Cheh, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013P001629
Record Dates: First submitted 2013-08-30; First posted 2013-09-06 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin group (Experimental): Healthy volunteers with QT genotype score in the highest or lowest quintile
  Interventions: Drug: Moxifloxacin 400mg once time
- Placebo group (Placebo Comparator): Healthy volunteers with QT genotype score in the highest or lowest quintile
  Interventions: Drug: Moxifloxacin 400mg once time

INTERVENTIONS:
Drug: Moxifloxacin 400mg once time
  Other Names: Avelox

SUMMARY:
The purpose of this study is to assess the ability of common genetic variants in aggregate to predict drug-induced QT prolongation in healthy subjects using moxifloxacin.

DETAILED DESCRIPTION:
I. Background and Significance A. Historical Background and Scientific Basis The most common cause of withdrawal or restriction of drugs that are already on the market is prolongation of the QT interval, and the consequent, potentially fatal, arrhythmia, torsade de pointes1. First described in the 1960s with quinidine therapy2, torsade de pointes occurs most commonly with antiarrhythmics3, although sudden cardiac death risk is increased 270% with use of a non-cardiac QT-prolonging medication4.

The QT interval of the electrocardiogram reflects ventricular myocardial repolarization, and abnormalities in the duration of the QT interval are the most common indicator of abnormal repolarization. Although a number of hypotheses exist for how abnormal repolarization, and specifically QT prolongation, results in ventricular arrhythmias, the most consistent finding appears to be that during prolonged depolarization sodium channels recover from inactivation and reactivate, causing what are termed early afterdepolarizations. When combined with heterogeneity in repolarization as well, these early afterdepolarizations create a favorable myocardial substrate for reentry, resulting in propagation of intramyocardial reentry waves and torsade de pointes5.

Drug-induced QT prolongation is the number one barrier for new therapeutic agents making it to market. While a number of medications, environmental factors, and genetic factors have been associated with QT prolongation, our ability to predict on an individual basis who will develop QT prolongation, not to mention torsade de pointes, is limited.

A personalized genetic approach to toxicity prevention would be important because cardiotoxic drug response is not specific to a single class of drugs; risk prediction for arrhythmogenicity can be applied across medications used in a variety of conditions. Narrowly, this research can enable drugs with currently marginal risk/benefit profiles to be brought to market, sparing those at-risk and providing access to new therapies for those who are not. From a public health perspective, it will reduce potentially fatal toxicity and thus improve human health through identification of particular at-risk individuals.

B. Previous Studies In a meta-analysis of three prospective cohorts--Cardiovascular Health Study, the Framingham Heart Study, and the Rotterdam Study--in 13,685 white people of European descent as part of the QTGEN consortium, Newton-Cheh and colleagues identified common variant associations (p < 5x10-8) at five loci previously associated with QT interval: NOS1AP, KCNQ1, KCNE1, KCNH2, and SCN5A, as well as new associations in 5 other loci previously unrecognized to influence myocardial repolarization10. At these 10 loci, 14 independent variants explained 5.4 - 6.5% of the variation of the QT interval, which was more than is explained by sex or age, the strongest non-genetic clinical factors10. A QT genotype score based on these variants was associated with a 9.7 - 12.4ms longer QTc in the top quintile compared with the bottom quintile in the meta-analysis samples, which included heterogeneous age, risk factor and drug exposure profiles10-12. These effects were consistent in individuals of both European and African American ancestry. This QT score was independently validated in a Finnish population sample in which complete medication ascertainment enabled excluding those on QT-altering therapy, and in which the QT score was associated with a 15.6ms QT interval difference between the top and bottom quintiles13.

Moxifloxacin is well-suited to study drug-induced QT prolongation, as it is known to cause transient and mild QT prolongation. Compared to placebo, 400mg of oral moxifloxacin is associated with an approximately 10 msec increase in the heart rate-corrected QT interval14, 15. Despite this increase in QT interval, there is no reported increased risk of sudden death with oral administration of a single dose of moxifloxacin16, so it is a safe and well-validated drug to use in the study of cardiotoxic drug response in healthy human subjects. Moreover, it has been widely used by the pharmaceutical industry as a positive control as required by the FDA to demonstrate a sufficiently sensitive method to detect QT prolongation.

C. Rationale of Proposed Benefit of Research Drug-induced QT prolongation is a significant public health risk and a major barrier to drug development19-21. For example, cisapride, an esophageal motility agent used for gastro-esophageal reflux, may have resulted in more than 80 deaths before it was pulled from the market22. In addition to identification of culprit medications, there are also characteristics of the vulnerable patient, including female sex23, bradycardia24, hypokalemia25, and genetic predisposition by rare mutations3, 6, 26, that place certain individuals at higher risk of fatal arrhythmia. Identification of these at-risk individuals with the use of genetic markers would represent a critical advance toward safer pharmacotherapy7. The basis of this study is to expand the use of genetics beyond rare family mutations that predispose to risk of QT prolongation to large-scale screening of the general population by genotyping (assaying for specific variants) for relatively common polymorphisms that could increase risk of QT prolongation, and subsequent torsade de pointes.

II. Specific Aim We hypothesize that common genetic variants with intermediate effects on resting QT, when examined in aggregate, can identify a subgroup of individuals at risk of exaggerated prolongation of the QT interval in response to a QT-prolonging medication.

This hypothesis will be tested through the following specific aim:

To assess the ability of common genetic variants in aggregate to predict drug-induced QT prolongation in healthy subjects. We will recruit 80 healthy volunteers drawn from the top and bottom quintiles of a QT genotype score for assessment of QT response to moxifloxacin compared to placebo at the Massachusetts General Hospital (MGH).

III. Subject Selection A. Inclusion/Exclusion Criteria: Through a separate protocol, Dr. Newton-Cheh has recruited to date over 1000 healthy volunteers aged 18 to 40 with consent for re-contact on the basis of genotypes determined after an initial screening visit, all of whom have undergone DNA extraction. From the existing collection of 1000 subjects, approximately 75% are self-described European/Caucasian and 8% are African Americans. These are otherwise healthy individuals ages 18 and older. For this study, we will genotype 68 independent QT SNPs using the Sequenom genotyping array in the MGH Center for Human Genetic Research Sequenom core on these samples. The genotype score is the sum of the predicted effects on QT interval for each genotype. From the genotype score, we will determine the set of individuals who belong to the top or bottom quintile of QT genotype risk score to be eligible for our moxifloxacin study (see below for details of the genotype score calculation). Apparently healthy male and female volunteers of European and African American ancestry, between 18 and 50 years old, will be eligible if they are free of known cardiovascular, renal, hepatic disease, have no personal or family history of sudden cardiac death; use no prescribed or over-the-counter medications as well as recreational drugs; have no bradycardia (defined as resting heart rate < 50 bpm), conduction disease (QRS > 100ms) or QTc prolongation on electrocardiography (QTc > 500msec); and have a normal serum potassium (K>3.3) and magnesium (Mg>1.8), as well as renal and liver function tests. We will exclude woman who are nursing, pregnant or planning to become pregnant during the study period, counsel them on the importance of using birth control during the study period, and check a serum HCG on the screening visit. We estimate that 266 individuals (133 in the highest and lowest quintiles, respectively) will be eligible.

IV. Subject Enrollment

A. Methods of Enrollment and Procedures for Informed Consent:

See above for details of subject identification for enrollment. Eligible individuals will be invited to come in for a screening visit for the moxifloxacin study with a target enrollment of 40 in each genotype group. We plan to contact up to 266 individuals who are in the upper and lower quintiles of QT genotype score to come in for the screening visit. We anticipate inviting approximately 160 individuals for the screening visit, with a goal enrollment sample size of 80 individuals. These subjects will be contacted by phone about participation in this study, and then informed consent will be obtained on arrival for the screening visit, and verified at subsequent visits if they are eligible for the study protocol.

V. Study Protocol A. Data Collection: Subjects will be brought to the MGH Clinical Research Center for an initial screening visit in which eligibility criteria will be reviewed (with exclusion/inclusion as applicable), and they will be given an ECG recording. Eligible individuals for the study visits will be brought back later to the MGH Clinical Research Center on two separate days separated by at least one week (to ensure washout). On each visit, they will receive study drug (either 400 mg oral moxifloxacin or placebo) allocated by double blinded block randomization (by sex and genotype group separately) at 10AM in the fasting state (statistician will hold the randomization key; all other study personnel will be blinded until study closure). Women will be screened for pregnancy using a urine HCG at the time of both study visits. They will undergo 6 ECGs at time 0 and at 30 min intervals thereafter, in the seated position after at least 15 min rest using fixed electrode placement for a total of 6 hours following administration of study drug. At 2, 4 and 6 hours we will draw a blood sample for plasma moxifloxacin determination by mass spectrometry. All ECGs are uploaded to a research partition of the GE MUSE 7 ECG database of the Massachusetts General Hospital, and the 12 SL algorithm applied for interval measurement, as used in prior studies by our group. We will monitor the QT every 30 minutes throughout the protocol and will identify any subjects with marked QT prolongation. Any subject who has a QTc >500 ms will be kept in the HCRC for further observation, with the decision to either follow-up at the HCRC every morning until it is less than 500ms or be admitted to the hospital for telemetry based on the degree of prolongation and clinician's judgment.

B. Venipuncture: Venipuncture will be performed using standard techniques to obtain plasma for quantification of moxifloxacin levels. We will collect 10 mL of blood at 2hrs, 4hr and 6hrs after study drug administration (Total 30mL).

C. Genotyping: Genotyping will be performed by the Sequenom genotyping array in the MGH Center for Human Genetic Research Sequenom core on existing genomic DNA isolated in.

VI. Biostatistical Analysis:

QT Genotype Score. We plan to use a modification of the QT genotype score that has been previously established11, 12 and validated by us in a separate Finnish cohort13. The score is constructed using allele copy number multiplied by effect estimates From the genotype score, we will determine the set of individuals who belong to the top or bottom quintile of QT genotype risk score (of whom, we expect 75% (n=133 per quintile)) to be eligible for our moxifloxacin study, based on our prior pilot work. We will invite these individuals to come in for a screening visit (see above) for the moxifloxacin study with a target enrollment of 40 in each genotype group.

Outcome assessment: Any individual with sinus arrhythmia present in over 50% of ECGs during the two study visits will be dropped from analysis. ECGs with premature ventricular or atrial beats will be dropped from analysis (these are very uncommon in healthy volunteers). The QTc using Fridericia's heart rate correction (QTc = QT/3√RR) will be taken as the average of all eligible ECGs from each time point. The ΔQTc will be calculated as the difference in QTc from baseline (after study drug/placebo administration) for each time point. From the ΔQTc, the difference between the post-moxifloxacin and post-placebo ΔQTc will then be calculated at each time point (ΔΔQTc) as well. The mean ΔΔQTc from the 180-300 minute time points (which from our pilot work and published reports is expected to be 10 msec) will then be compared between the two genotype groups (top and bottom and quintile) using an unpaired t-test. We estimate that 40 people in each group will be needed to have adequate power to detect a clinically meaningful (6.3 msec) difference in QT-prolongation between the two groups based on our pilot data (Table 2). An increase of 6 msec after exposure to a drug compared to placebo is the threshold at which the FDA raises concern for the potential of a drug to cause torsade de pointes and is thus clinically significant.

Secondary analyses. We plan to perform three secondary analyses. First, we will examine the influence of single SNPs of stronger effect on QT response to moxifloxacin. As power calculations, and study enrollment are based on the aggregated genotype score, we expect these secondary analyses to be underpowered. Second, if we observe a significant difference in QT response between top and bottom quintiles of QT genotype score, we will examine the influence of deciles on observed results comparing the 9th (80-90%ile) and 10th deciles (>90%ile) of score to the bottom decile or quintile, although given the composite nature of the genotype score and additive nature of the variants, we do not expect a threshold effect. Lastly, we will determine the impact of baseline QTc on QT response and test whether additional adjustment for baseline QTc alters any observed effect of genotype score on QT response to moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Genotype in the highest and lowest quintiles of genetic predictors of QT interval duration
* Able to swallow pills

Exclusion Criteria:

* Inability to provide informed consent
* Prior known cardiovascular, renal, hepatic disease
* Personal or family history of sudden cardiac death
* Current use of prescribed or over-the-counter medications as well as recreational drugs
* Resting bradycardia (defined as resting heart rate < 50 bpm)
* Conduction disease (QRS > 100ms)
* QTc prolongation on electrocardiography (QTc > 500msec)
* Abnormal potassium or magnesium serum level
* Abnormal renal or liver function tests
* Women who are nursing, pregnant or planning to become pregnant during the study period
* Tendon disorder or rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
QT interval duration | 6 Hours
  We will measure the QT interval on ECG up to 6 hours after administration of moxifloxacin or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Newton-Cheh, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States